CLINICAL TRIAL: NCT06587659
Title: Accelerated Image-Guided Robotically Delivered Transcranial Magnetic Stimulation for Combat PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Trauma Research and Combat Casualty Care Collaborative (Unknown)
Responsible Party: Principal Investigator, Felipe S. Salinas, Ph.D., Assistant Professor-Research, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000504
Record Dates: First submitted 2024-05-28; First posted 2024-09-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Nonrandomized, open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- IR-TMS to the right DLPFC (Experimental): IR-TMS will be delivered to the right DLPFC using connectivity-based, image-guided aiming with the IR-TMS coil positioned using a robotic arm. In this arm, active IR-TMS will be delivered using a theta burst stimulation protocol (i.e. 1,800 pulses/session), 4 sessions per day, 5 days/week, for 2 weeks.
  Interventions: Device: Transcranial Magnetic Stimulation; Device: Robotic Arm

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The MagPro R30 is an advanced, high performance magnetic stimulator designed primarily for non-invasive clinical use. The non-invasive brain stimulation system will be used to deliver active repetitive electromagnetic pulses in this research study's treatment of post-traumatic stress disorder.
  Other Names: TMS
Device: Robotic Arm — This robotic system is based on a commercially available collaborative robot. The robot is mounted on a cart which holds the robot controller and the TMS power supply and pulse-generation computer. The robotic system will be used for TMS coil positioning/targeting.

SUMMARY:
Posttraumatic stress disorder (PTSD) among military service members and veterans is as high as 32% and is the third most service-connected disability, resulting in over $1.5 billion in direct costs over a five-year period. According to Clinical Practice Guidelines, strong evidence exists for psychotherapies, such as prolonged exposure (PE) for PTSD. However, psychotherapies are often met with high drop-out rates, treatment non-compliance, and emotional stress due to trauma recall. A successful approach to reduce drop-out rates and maintain efficacy is to compress psychotherapy into daily, day-long PE sessions. Yet another deficit exists regarding the feasibility of this approach outside of residential treatment facilities, which are typically reserved for the most extreme cases. The newest study from the our team aimed to augment PE residential treatment with a neuromodulatory treatment: image-guided, robot-navigated transcranial magnetic stimulation (IR-TMS). Along with the PE-focused intensive inpatient program (IIP-PE), participants received IR-TMS targeting the right dorsolateral prefrontal cortex (DLPFC) daily for 20 consecutive days. Results demonstrated superiority of the combined IIP-PE/IR-TMS approach, compared to IIP-PE and a sham condition. However, it is not yet established whether a standalone IR-TMS approach will achieve similar results. Our goal is to implement an open-label trial of IR-TMS for PTSD, in which veterans and active-duty service members with PTSD will receive accelerated IR-TMS throughout a 2-week timeframe. Results will be used as a foundation for future extramural funding to scale-up the stand alone IR-TMS intervention for PTSD treatments.

DETAILED DESCRIPTION:
We propose an open-label, 2-week trial of IR-TMS targeting the right, anterior dorsolateral prefrontal cortex (R-antDLPFC) in 30 PTSD participants. We will recruit Active-Duty Service Members and Veterans with combat PTSD, as determined by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5). Participants will be encouraged to complete as many IR-TMS sessions throughout a 2-week time period, with a maximum of 4 sessions per day. Treatments will be neuro-navigated and adapted for an accelerated TMS treatment schedule. Post-Treatment and durability of this treatment effect will be examined throughout the 1-month and 3-month FU assessments. Findings from this open-label trial of IR-TMS for PTSD will serve as preliminary data for a larger randomized clinical trial to further identify the stand-alone effects of IR-TMS versus a sham condition.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18 and 70 years
2. meet diagnostic criteria for PTSD on the CAPS-5
3. able to attend all clinic appointments
4. fluent in English

Exclusion Criteria:

1. a documented diagnostic history of bipolar disorder, schizophrenia or schizoaffective disorder or a psychiatric hospitalization in the last 12 months
2. significant cognitive impairment determined by inability to comprehend screening assessment
3. psychiatric problems and/or high suicide risk warranting immediate intervention, as assessed with the PHQ-9 (Item #9)
4. currently meeting a psychiatric diagnosis of alcohol and/or substance abuse that would prevent the participant from engaging in therapy
5. any history or signs of serious medical or neurological illness including seizure disorders
6. history of traumatic brain injury (TBI) with loss of consciousness for 20 minutes or more
7. females will be excluded if they are pregnant
8. any history or signs of metal objects deemed unsafe for MRI or that may adversely affect image quality of the brain region (e.g. surgical clips, cardiac pacemakers, metal implants, etc.) in the body at the time of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Severity as Measured by the PTSD Checklist (PCL-5) | Baseline to two weeks (the conclusion of IR-TMS treatment)
  PTSD Checklist for DSM-5 (PCL-5) has excellent psychometric characteristics for screening and as a secondary indicator of PTSD symptom severity. The PCL-5 is a 20-item self-report measure, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. Scoring is based on how much the participant has been bothered by the symptoms in the past month on a scale from "0 = not at all" to "4 = extremely." Items are summed to provide a total severity score (range = 0-80). If the participant scores above 33 in total, it is probable that they have PTSD. A clinically significant change in the PCL-5 is a 10-20 point change in the total symptom severity score. A 5-10 point change is considered a reliable change, meaning it is not due to chance.

SECONDARY OUTCOMES:
Change in PTSD Severity as Measured by the PTSD Checklist (PCL-5) | Baseline to one week (mid IR-TMS treatment)
  PTSD Checklist for DSM-5 (PCL-5) has excellent psychometric characteristics for screening and as a secondary indicator of PTSD symptom severity. The PCL-5 is a 20-item self-report measure, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. Scoring is based on how much the participant has been bothered by the symptoms in the past month on a scale from "0 = not at all" to "4 = extremely." Items are summed to provide a total severity score (range = 0-80). If the participant scores above 33 in total, it is probable that they have PTSD. A clinically significant change in the PCL-5 is a 10-20 point change in the total symptom severity score. A 5-10 point change is considered a reliable change, meaning it is not due to chance.
Change in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9) | Baseline to one week (mid IR-TMS treatment)
  The Participant Health Questionnaire-9 (PHQ-9) is a widely used and well-validated instrument for measuring the severity of depressive symptoms. It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders; these 9 items correspond to the DSM diagnostic criteria for Major Depressive Disorder. Respondents rate the frequency with which they have been bothered by depressive symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"); PHQ-9 scores range from 0 to 27. Scores reflect no significant depressive symptoms (0-4), mild depressive symptoms (5-9), moderate depressive symptoms (10-14), moderately severe depressive symptoms (15-19), and severe depressive symptoms (20-27). A 5-point change is clinically significant. A score of less than 10 suggests a partial response, and a score of less than 5 represents remission.
Change in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9) | Baseline to two weeks (the conclusion of IR-TMS treatment)
  The Participant Health Questionnaire-9 (PHQ-9) is a widely used and well-validated instrument for measuring the severity of depressive symptoms. It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders; these 9 items correspond to the DSM diagnostic criteria for Major Depressive Disorder. Respondents rate the frequency with which they have been bothered by depressive symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"); PHQ-9 scores range from 0 to 27. Scores reflect no significant depressive symptoms (0-4), mild depressive symptoms (5-9), moderate depressive symptoms (10-14), moderately severe depressive symptoms (15-19), and severe depressive symptoms (20-27). A 5-point change is clinically significant. A score of less than 10 suggests a partial response, and a score of less than 5 represents remission.
Change in PTSD Severity as Measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline to six weeks (4 weeks post IR-TMS treatment)
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a structured diagnostic interview and gold standard for assessing PTSD. The scale also assesses social and occupational functioning, dissociation, and the validity of symptom reports. Symptom severity ratings combine information about symptom frequency and intensity obtained by the interviewer. CAPS-5 scores range from 0 to 80 with higher scores indicating greater PTSD symptom severity. A clinically significant change in the CAPS-5 is a score of 8 or less. A reliable change in CAPS-5 scores is a change of 13 or more.
Change in PTSD Severity as Measured by the PTSD Checklist (PCL-5) | Baseline to six weeks (4 weeks post IR-TMS treatment)
  PTSD Checklist for DSM-5 (PCL-5) has excellent psychometric characteristics for screening and as a secondary indicator of PTSD symptom severity. The PCL-5 is a 20-item self-report measure, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. Scoring is based on how much the participant has been bothered by the symptoms in the past month on a scale from "0 = not at all" to "4 = extremely." Items are summed to provide a total severity score (range = 0-80). If the participant scores above 33 in total, it is probable that they have PTSD. A clinically significant change in the PCL-5 is a 10-20 point change in the total symptom severity score. A 5-10 point change is considered a reliable change, meaning it is not due to chance.
Change in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9) | Baseline to six weeks (4 weeks post IR-TMS treatment)
  The Participant Health Questionnaire-9 (PHQ-9) is a widely used and well-validated instrument for measuring the severity of depressive symptoms. It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders; these 9 items correspond to the DSM diagnostic criteria for Major Depressive Disorder. Respondents rate the frequency with which they have been bothered by depressive symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"); PHQ-9 scores range from 0 to 27. Scores reflect no significant depressive symptoms (0-4), mild depressive symptoms (5-9), moderate depressive symptoms (10-14), moderately severe depressive symptoms (15-19), and severe depressive symptoms (20-27). A 5-point change is clinically significant. A score of less than 10 suggests a partial response, and a score of less than 5 represents remission.
Change in PTSD Severity as Measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline to fourteen weeks (12 weeks post IR-TMS treatment)
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a structured diagnostic interview and gold standard for assessing PTSD. The scale also assesses social and occupational functioning, dissociation, and the validity of symptom reports. Symptom severity ratings combine information about symptom frequency and intensity obtained by the interviewer. CAPS-5 scores range from 0 to 80 with higher scores indicating greater PTSD symptom severity. A clinically significant change in the CAPS-5 is a score of 8 or less. A reliable change in CAPS-5 scores is a change of 13 or more.
Change in PTSD Severity as Measured by the PTSD Checklist (PCL-5) | Baseline to fourteen weeks (12 weeks post IR-TMS treatment)
  PTSD Checklist for DSM-5 (PCL-5) has excellent psychometric characteristics for screening and as a secondary indicator of PTSD symptom severity. The PCL-5 is a 20-item self-report measure, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. Scoring is based on how much the participant has been bothered by the symptoms in the past month on a scale from "0 = not at all" to "4 = extremely." Items are summed to provide a total severity score (range = 0-80). If the participant scores above 33 in total, it is probable that they have PTSD. A clinically significant change in the PCL-5 is a 10-20 point change in the total symptom severity score. A 5-10 point change is considered a reliable change, meaning it is not due to chance.
Change in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9) | Baseline to fourteen weeks (12 weeks post IR-TMS treatment)
  The Participant Health Questionnaire-9 (PHQ-9) is a widely used and well-validated instrument for measuring the severity of depressive symptoms. It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders; these 9 items correspond to the DSM diagnostic criteria for Major Depressive Disorder. Respondents rate the frequency with which they have been bothered by depressive symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"); PHQ-9 scores range from 0 to 27. Scores reflect no significant depressive symptoms (0-4), mild depressive symptoms (5-9), moderate depressive symptoms (10-14), moderately severe depressive symptoms (15-19), and severe depressive symptoms (20-27). A 5-point change is clinically significant. A score of less than 10 suggests a partial response, and a score of less than 5 represents remission.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe S Salinas, Ph.D., Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- Research Imaging Institute, San Antoio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD may be shared with other researchers who have been granted a data sharing agreement with the research team and/or the study sponsor. A description of the types of data collected for each individual will be provided. De-identified IPD will consist of symptom scores for the PCL-5, PHQ-9 , and CAPS-5 assessments will be shared for each time point in which they are (respectively) acquired.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be made available at the end of the study (anticipated July 2025) and will be made available to the public for at least 2 years after study completion (anticipated July 2027).
Access Criteria: De-identified IPD may be shared with other researchers who have been granted a data sharing agreement with the research team and/or the study sponsor. A description of the types of data collected for each individual will be provided. De-identified IPD will consist of symptom scores for the PCL-5, PHQ-9 , and CAPS-5 assessments will be shared for each time point in which they are (respectively) acquired. Data sharing requests must be submitted to the study team. If granted access, the requestor will be sent a digital link to a shared repository folder (maintained by the study PI).